CLINICAL TRIAL: NCT03203603
Title: Vitamin C to Decrease the Effects of Smoking in Pregnancy on Infant Lung Function (VCSIP): Follow-up of a Randomized Trial
Brief Title: VCSIP Follow-up Study
Acronym: VCSIPRenewal
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Indiana University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Cynthia McEvoy, MD, MCR, Oregon Health and Science University
Other Study IDs: VCSIP-Renewal
Record Dates: First submitted 2017-03-28; First posted 2017-06-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Asthma; Pulmonary Function; Wheezing; In Utero Nicotine
Keywords: asthma; pulmonary function testing; wheeze; vitamin C; antioxidants; forced expiratory flows
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — buccal swabs, hair, blood and urine will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Offspring of smokers who got vitamin C: Offspring of pregnant smokers randomized to vitamin C during the initial randomized portion of the VCSIP study
  Interventions: Other: No active intervention
- Offspring of smokers who got placebo: Offspring of pregnant smokers randomized to placebo during the initial randomized portion of the VCSIP study
  Interventions: Other: No active intervention
- Offspring of pregnant non-smokers: Offspring of pregnant non-smokers who were followed in a similar fashion during pregnancy as the randomized pregnant smokers
  Interventions: Other: No active intervention

INTERVENTIONS:
Other: No active intervention — This is a follow-up of a randomized trial. No active intervention is being given in the follow-up.

SUMMARY:
The overall aims of this protocol are to determine whether prenatal supplementation with vitamin C to pregnant smokers can improve pulmonary function and decrease wheeze at 5 years of age in their offspring. This is a continuation of the VCSIP trial, to follow the offspring through 5 years of age. The hypothesis for this protocol is an extension of the VCSIP trial that supplemental vitamin C in pregnant smokers can significantly improve their children's PFTs and decrease the incidence of wheeze.

DETAILED DESCRIPTION:
The overall aims of this protocol are to determine whether prenatal supplementation with vitamin C to pregnant smokers can improve pulmonary function and decrease wheeze at 5 years of age in their offspring. This is a continuation of the VCSIP trial, to follow the offspring through 5 years of age. The hypothesis for this protocol is an extension of the VCSIP trial that supplemental vitamin C in pregnant smokers can significantly improve their children's PFTs and decrease the incidence of wheeze. The reasons for this protocol are to follow the children born to mothers randomized in the VCSIP to the age of 5 to differentiate the patients with transient versus recurrent wheeze (and therefore more likely to develop asthma); to determine if early protective effects of vitamin C are sustained to this older age; and to continue to collect biologic samples from the children for future mechanistic studies of vitamin C action.

The primary aim of this study is to demonstrate improved pulmonary function at 5 years of age in the offspring of pregnant smokers randomized to vitamin C (500 mg/day) versus placebo. The investigators hypothesize that vitamin C supplementation in pregnancy will block the adverse effects of maternal smoking on offspring pulmonary function measured at 5 years of age by spirometry. Impulse oscillometry (IOS) will also be used at 3-5 years of age to assess pulmonary function.

Specific Aim 2 (Secondary Outcome): The secondary aim of this study is to demonstrate a decreased incidence of wheeze at 5 years of age in offspring of pregnant smokers randomized to vitamin C (500 mg/day) versus placebo. The investigators hypothesize that vitamin C supplementation during pregnancy will decrease the incidence of wheeze at 5 years of age in offspring of smokers. Respiratory health will be assessed by quarterly validated respiratory questionnaires and clinician report.

ELIGIBILITY:
Inclusion Criteria:

* Women and their offspring randomized to vitamin C versus placebo during pregnancy as well as pregnant nonsmokers and their offspring enrolled as the reference group in the current RCT.

Exclusion Criteria:

* Patients specifically withdrawing consent.

Ages: 6 Months to 4 Years | Sex: All
Age Groups: Child
Study Population: This is a follow up of NCT01723696. In that study, pregnant smokers were recruited at obstetric clinics delivering at OHSU, PeaceHealth Southwest Washington Medical Center in Vancouver, Washington or Indiana University in Indianapolis, Indiana. We are now following the offspring of those pregnant smokers (and control group non-smokers).
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Improved pulmonary function, spirometry | 5 years of age
  The primary aim of this study is to demonstrate improved pulmonary function at 5 years of age in the offspring of pregnant smokers randomized to vitamin C 500 mg/day versus placebo.

SECONDARY OUTCOMES:
Decreased incidence of wheeze | 5 years of age
  The secondary aim of this study is to demonstrate a decreased incidence of wheeze at 5 year of age in offspring of pregnant smokers randomized to vitamin C (500 mg/day) versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Cindy McEvoy, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McEvoy CT, Schilling D, Clay N, Jackson K, Go MD, Spitale P, Bunten C, Leiva M, Gonzales D, Hollister-Smith J, Durand M, Frei B, Buist AS, Peters D, Morris CD, Spindel ER. Vitamin C supplementation for pregnant smoking women and pulmonary function in their newborn infants: a randomized clinical trial. JAMA. 2014 May;311(20):2074-82. doi: 10.1001/jama.2014.5217. PMID 24838476
- [Derived] Shorey-Kendrick LE, McEvoy CT, Milner K, Harris J, Brownsberger J, Tepper RS, Park B, Gao L, Vu A, Morris CD, Thompson EE, Ober C, Spindel ER. Vitamin C supplementation to pregnant smokers alters asthma- and allergy-associated CpGs in child buccal DNA at 5 years of age. Clin Epigenetics. 2025 Oct 3;17(1):155. doi: 10.1186/s13148-025-01965-2. PMID 41044653
- [Derived] Shorey-Kendrick LE, McEvoy CT, Milner K, Harris J, Brownsberger J, Tepper RS, Park B, Gao L, Vu A, Morris CD, Spindel ER. Improvements in lung function following vitamin C supplementation to pregnant smokers are associated with buccal DNA methylation at 5 years of age. Clin Epigenetics. 2024 Feb 27;16(1):35. doi: 10.1186/s13148-024-01644-8. PMID 38413986
- [Derived] McEvoy CT, Shorey-Kendrick LE, Milner K, Harris J, Vuylsteke B, Cunningham M, Tiller C, Stewart J, Schilling D, Brownsberger J, Titus H, MacDonald KD, Gonzales D, Vu A, Park BS, Spindel ER, Morris CD, Tepper RS. Effect of Vitamin C Supplementation for Pregnant Smokers on Offspring Airway Function and Wheeze at Age 5 Years: Follow-up of a Randomized Clinical Trial. JAMA Pediatr. 2023 Jan 1;177(1):16-24. doi: 10.1001/jamapediatrics.2022.4401. PMID 36409489